CLINICAL TRIAL: NCT04366193
Title: Validation of a High-resolution Oximeter Using a Cloud-based Algorithm to Diagnose Obstructive Sleep Apnea
Brief Title: High-resolution Oximetry to Diagnose Obstructive Sleep Apnea
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Geraldo Lorenzi Filho, Associate Professor, University of Sao Paulo General Hospital
Other Study IDs: 3767871
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Sleep Apnea
Keywords: sleep apnea; home sleep test; oximetry
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Oximetry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Oximetry — Validation of a high-resolution wireless oximeter for OSA diagnosis comparing with a well established and validated method (home sleep test).

SUMMARY:
The aim of this study was to compare an overnight digital monitoring device (ODM) with home sleep apnea testing (HSAT) using respiratory flow and effort parameters in a large population sample, who were in a waiting list for Polysomnography (PSG).

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) is extremely common has prompted the popularization of home sleep test (HST). HST record a limited number of respiratory signals, provide a more comfortable testing option to the patient at a lower cost. HST has a performance as good as PSG among patients with suspected OSA and no significant co-morbidities.

Our study was designed to investigate the performance of a simple solution that consists of a high-resolution wireless oximeter with a built-in accelerometer linked to a smartphone application and automated cloud algorithm for detection of oxygen desaturation, described herein as Overnight Digital Monitoring (ODM) (BilogixTM). We will compare the results of ODM with HST performed by ApneaLink Air by Resmed®.

We have already compared ODM to PSG with excellent results in a prior study and intend to see the results in uncontrolled environment (home) .

Population: Men and women from the São Paulo Department of Health, who are awaiting examination for diagnosis of OSAS.We intend to compare the ODM with the HST. Patients with indication for CPAP titration will be excluded. The participants will wear a wireless oximeter (Oxistar, Biologix Sistemas Ltda., Brazil) with a built-in accelerometer on a finger of the same hand as the HST oximeter and we will compare both methods for diagnosing OSA.

All HST studies will be scored by 2 independent certified technicians blinded to the ODM results. Hypopnea will be defined as a peak signal excursion drop by ≥ 30% of pre-event baseline nasal pressure signal lasting ≥ 10 sec. Hypopneas will be scored according the acceptable AASM criteria for hypopnea (≥ 4% reduction in SpO2). Mild, moderate and severe OSA will be defined according to the current standards (5 ≤ AHI <15; 15 ≤ AHI <30 and AHI ≥30 events/h, respectively).ODI results from ODM will be expressed as the number of desaturations per recording time and will be automatically analyzed at the cloud. In order to compare with TST-AHI4%, ODM will be matched using 4% desaturation criteria (ODM-ODI4%, respectively).

ELIGIBILITY:
Inclusion Criteria:

* Adult ambulatory patients who are in a waiting list for polysomnography that are able to properly place the oximeter and home sleep test at home

Exclusion Criteria:

* patients under treatment for OSA

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult ambulatory patients who are in a waiting list for polysomnography
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-12-12 (Actual); Primary Completion 2020-04-16 (Actual); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of high-resolution oximetry for OSA | single night
  Accuracy will be tested against home sleep test using ROC, sensitivity and specificity

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep Laboratory, Heart Institute, Pulmonary Division, Hospital das Clínicas da Universidade de São Paulo, São Paulo, Brazil